CLINICAL TRIAL: NCT00021047
Title: A Phase I/II Trial of Epirubicin, Carboplatin & Capecitabine in Adult Cancer Patients
Brief Title: Epirubicin, Carboplatin, and Capecitabine in Treating Patients With Unresectable Locally Advanced, Metastatic, or Recurrent Solid Tumor
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 010172; NCI-01-C-0172; MB-NAVY-00-07; MB-NAVY-B01-008; CDR0000068741; NCT00015743 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Esophageal Cancer; Extrahepatic Bile Duct Cancer; Gastric Cancer; Head and Neck Cancer; Liver Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV gastric cancer; recurrent gastric cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; unspecified adult solid tumor, protocol specific; untreated metastatic squamous neck cancer with occult primary; recurrent metastatic squamous neck cancer with occult primary; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV basal cell carcinoma of the lip; stage IV verrucous carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent verrucous carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; stage IV squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; stage IV salivary gland cancer
MeSH Terms: conditions — Esophageal Neoplasms; Bile Duct Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms; Liver Neoplasms; Carcinoma, Hepatocellular; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms | interventions — Capecitabine; Carboplatin; Epirubicin

INTERVENTIONS:
Drug: capecitabine
Drug: carboplatin
Drug: epirubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combining epirubicin, carboplatin, and capecitabine in treating patients who have unresectable locally advanced, metastatic, or recurrent solid tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and the recommended phase II dose of capecitabine administered with epirubicin and carboplatin in patients with unresectable locally advanced, metastatic, or recurrent solid tumors.
* Determine the toxic effects of this regimen in these patients.
* Determine the pharmacokinetics (PK) of capecitabine and correlate these PK parameters with clinical toxicity of this regimen in these patients.
* Correlate end-of-infusion levels of epirubicin and its metabolites with epirubicin dose and clinical toxicity of this regimen in these patients.
* Determine the possible correlation between polymorphisms in the promoter region of the thymidylate synthase gene with clinical toxicity of this regimen in these patients.
* Determine the antitumor activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study of capecitabine.

Patients receive epirubicin IV over 2 hours and carboplatin IV over 30 minutes on day 1 and oral capecitabine twice daily on days 2-5, 8-12, and 15-19. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 24 additional patients are treated at the recommended phase II dose.

PROJECTED ACCRUAL: A total of 3-45 patients (24 patients for phase II) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor

  * Progressive disease on standard therapy, including:

    * Locally advanced, unresectable primary or recurrent tumor OR
    * Metastatic disease
* Previously untreated metastatic cancer for which study regimen represents reasonable initial chemotherapy with palliative intent (e.g., metastatic gastric cancer, hepatobiliary cancer, or cancers for which no effective standard therapy exists) allowed
* Phase II portion:

  * Diagnosis of cancer of the upper aerodigestive tract (head and neck, esophagus, stomach, or hepatobiliary)
  * No potential curative treatment options including surgery, radiotherapy, chemoradiotherapy, or combination chemotherapy
  * No leukemia or lymphoma
  * No primary CNS malignancies or CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST and ALT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.6 mg/dL

Cardiovascular:

* LVEF at least 50%
* No symptomatic congestive heart failure
* No unstable angina
* No cardiac arrhythmia

Other:

* No serious concurrent medical illness that would preclude study participation
* No active infections requiring IV antibiotic therapy
* No history of allergy to platinum compounds, mannitol, or antiemetics used with study drugs
* No history of severe intolerance to fluorouracil
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* More than 4 weeks since prior immunotherapy and recovered

Chemotherapy:

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy (at least 6 weeks for nitrosoureas or mitomycin) and recovered
* No prior cumulative doxorubicin dose of more than 300 mg/m2

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 2 weeks since prior radiotherapy and recovered
* At least 8 weeks since prior strontium chloride Sr 89

Surgery:

* See Disease Characteristics
* Recovered from prior surgery

Other:

* At least 4 weeks since prior sorivudine or brivudine
* No concurrent sorivudine or brivudine
* No concurrent cimetidine
* No concurrent antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-07; Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian P. Monahan, MD, FACP — National Cancer Institute (NCI); Eva Szabo, MD, Study Chair — National Cancer Institute (NCI)
Locations (3):
- United States (3):
  - Center for Cancer Research, Bethesda, Maryland
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia